CLINICAL TRIAL: NCT00807144
Title: A Phase-IV Study Comparing Standard Release Tacrolimus (Prograf) vs Prolonged-release Tacrolimus (Advagraf) Monotherapy as Maintenance Immunosuppression After Induction With Alemtuzumab in Kidney Transplantation
Brief Title: Standard Versus Prolonged-release Tacrolimus Monotherapy After Alemtuzumab Induction in Kidney Transplantation
Acronym: TAESR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICKTI08TX02; 2008-000889-22 (EudraCT Number)
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: End-stage Renal Failure; Graft Rejection
Keywords: Kidney transplant; Rejection; Adherence; Quality of life
MeSH Terms: conditions — Kidney Failure, Chronic; Rejection, Psychology | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged-Release Tacrolimus (Experimental): Transplant maintenance immunosuppression with Prolonged-release Tacrolimus monotherapy
  Interventions: Drug: Kidney transplant maintenance immunosuppression
- Standard-Release tacrolimus (Active Comparator): Transplant maintenance immunosuppression with Standard-release Tacrolimus monotherapy
  Interventions: Drug: Tacrolimus (Kidney transplant maintenance immunosuppression)

INTERVENTIONS:
Drug: Tacrolimus (Kidney transplant maintenance immunosuppression) — Standard-release Tacrolimus 1 to 20mg daily in two divided doses to maintain trough drug levels 6-9ng/ml
  Other Names: Prograf
  Arms: Standard-Release tacrolimus
Drug: Kidney transplant maintenance immunosuppression — Prolonged-release Tacrolimus 1 to 20mg daily in a single am dose adjusted to trough drug levels 6-9ng/ml
  Other Names: Advagraf
  Arms: Prolonged-Release Tacrolimus

SUMMARY:
The current anti-rejection drug regime for kidney transplant recipients in use at the West London Renal & Transplant Centre (WLRaTC) consists of induction therapy with the very potent monoclonal antibody Campath 1-H (Alemtuzumab) followed by long-term maintenance with the Calcineurin inhibitor Tacrolimus

The recent development (and licensing in the UK) of an extended-release, once daily formulation of Tacrolimus holds out the promise of simpler drug regimes for our patients. In the context of our current successful use of Tacrolimus monotherapy maintenance after Campath 1-H induction, the extended-release Tacrolimus formulation will enable us to offer a regime where the only long-term immunosuppressive treatment that most of our patients need will be a single drug, taken once a day.

The investigators wish to assess the efficacy of such a regime in a structured comparison with our current protocol.

DETAILED DESCRIPTION:
1. Purpose of Study:

   The current immunosuppressive regime used as anti-rejection therapy after kidney transplantation in the West London Renal & Transplant Centre at Imperial College Healthcare NHS Trust consists of induction therapy with Campath 1-H(Alemtuzumab) and a 1 week course of steroids followed by maintenance mono-therapy with standard-release (twice daily) Tacrolimus (Prograf). This study is designed to compare the costs and outcomes of this regime with one in which extended-release (once daily) Tacrolimus (Advagraf) is used in place of the standard-release Tacrolimus.
2. Study Type: Phase IV
3. Study Design: Prospective, randomised, controlled, open study. Patients will be randomized 1:1 between the standard and extended-release Tacrolimus arms.

   Study entry will be stratified by live donor vs deceased donor transplants. The total recruitment target is 100 patients (50 standard release/50 extended release).
4. Study Description:

Patients will be randomised to receive either Prograf or Advagraf prior to transplantation.

Other than through the taking of extra blood samples at the time of routine clinical visits, participants will receive identical in-patient and out-patient management to patients undergoing kidney transplantation under our standard protocol.

Patients in the study will be asked to complete a short Health-Related Quality of Life questionnaire (SF-36) before transplantation and at 1 year post transplant. They will also be asked to complete a Medication Adherence Rating Score at 3, 6, and 12 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Live donor kidney transplant recipients
* heart-beating-Deceased donor kidney transplant recipients
* Patients suitable for induction therapy with Alemtuzumab

Exclusion Criteria:

* Recipients of Non-heart-beating deceased donor kidney transplants
* Recipients of simultaneous kidney/pancreas transplants
* ABO incompatible/desensitized transplant recipients
* Positive flow cross-match/desensitized transplant recipients
* Patients with heavy prior exposure to myelosuppressive therapy
* Patients with previous malignancy
* Patients with HIV,Hepatitis-C, or Hepatitis-B infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam G McLean, MA DPhil, Principal Investigator — Imperial College Kidney & Transplant Institute
Locations (1):
- West London Renal & Transplant Centre, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Conference abstract — https://atcmeetingabstracts.com/abstract/1-year-outcomes-of-a-prospective-open-label-randomized-controlled-trial-of-standard-vs-extended-release-tacrolimus-as-maintenance-monotherapy-in-kidney-transplantation-after-alemtuzumab-induction-w

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended Release Tacrolimus: Transplant maintenance immunosuppression with Prolonged-release Tacrolimus monotherapy
  Kidney transplant maintenance immunosuppression: Prolonged-release Tacrolimus 1 to 20mg daily in a single am dose adjusted to trough drug levels 6-9ng/ml
- Standard Release Tacrolimus: Transplant maintenance immunosuppression with Standard-release Tacrolimus monotherapy
  Tacrolimus (Kidney transplant maintenance immunosuppression): Standard-release Tacrolimus 1 to 20mg daily in two divided doses to maintain trough drug levels 6-9ng/ml
Period: Overall Study
Arm/Group | Extended Release Tacrolimus | Standard Release Tacrolimus
Started | 52 | 50
Completed | 52 | 49
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Release Tacrolimus | Standard Release Tacrolimus | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (15.8) | 51.5 (14.04) | 52.3 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 39 | 37 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Afro Carribean | 4 | 6 | 10
  Asian | 9 | 11 | 20
  Caucasian | 36 | 30 | 66
  Other | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 52 | 50 | 102

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival With a Functioning Graft
Time Frame: One year post kidney transplantation
Measure: Number; unit: percent of participants
Arm/Group | Extended Release Tacrolimus | Standard Release Tacrolimus
Number analyzed (Participants) | 52 | 50
percent of participants | 92.3 | 96
Statistical Analysis 1: Comparison: Extended Release Tacrolimus vs Standard Release Tacrolimus; Test type: Superiority; p = 0.26, Log Rank

2. Secondary Outcome: Rejection-free Patient Survival With a Functioning Graft
Time Frame: One and two years post kidney transplantation
Measure: Number; unit: percent of participants
Arm/Group | Extended Release Tacrolimus | Standard Release Tacrolimus
Number analyzed (Participants) | 52 | 50
percent of participants
  year 1 | 86 | 84
  year 2 | 83.4 | 80.1
Statistical Analysis 1: Comparison: Extended Release Tacrolimus vs Standard Release Tacrolimus; Year 1; Test type: Superiority; p = 0.48, Log Rank
Statistical Analysis 2: Comparison: Extended Release Tacrolimus vs Standard Release Tacrolimus; Year 2; Test type: Superiority; p = 0.75, Log Rank

3. Secondary Outcome: Patient-reported Quality of Life, and Medication Adherence
Time Frame: 3,6,& 12 months post kidney transplant
Population: Data not collected
Arm/Group | Extended Release Tacrolimus | Standard Release Tacrolimus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Extended Release Tacrolimus | Standard Release Tacrolimus
All-Cause Mortality (participants affected / at risk) | 4/52 | 2/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 1/50
Other Adverse Events (participants affected / at risk) | 8/52 | 9/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Tacrolimus (N=52) | Standard Release Tacrolimus (N=50)
Liver failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release Tacrolimus (N=52) | Standard Release Tacrolimus (N=50)
Any rejection symptom (General disorders) | 8 (8) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes